CLINICAL TRIAL: NCT00096408
Title: LACE - Laparoscopic Approach to Cancer of the Endometrium: An International Multicenter Randomized Phase 3 Clinical Trial
Brief Title: Laparoscopic Approach to Cancer of the Endometrium
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Queensland Centre for Gynaecological Cancer (Other Government)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry); Tyco Healthcare Group (Industry); Gynetech (Industry); Queensland Government - Smart Health Research Grant (Unknown); National Health and Medical Research Council, Australia (Other); Cancer Council Queensland (Other); Cancer Council New South Wales (Other); Cancer Council Victoria (Other); Cancer Council Western Australia (Unknown); Cancer Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LACE001
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Endometrial Cancer
Keywords: Endometrial; Endometrium; Uterus; Cancer; Carcinoma; Adenocarcinoma; Stage 1; Hysterectomy; Laparoscopy; Abdominal; Total; Surgery; Quality of Life; Disease-free survival
MeSH Terms: conditions — Endometrial Neoplasms; Neoplasms; Carcinoma; Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Total Abdominal Hysterectomy
  Interventions: Procedure: Total Abdominal Hysterectomy
- 2 (Experimental): Total Laparoscopic Hysterectomy
  Interventions: Procedure: Total Laparoscopic Hysterectomy

INTERVENTIONS:
Procedure: Total Abdominal Hysterectomy — For patients with clinical stage I disease, removal of the uterus and both tubes and ovaries are considered current standard treatment in Australia.
  Other Names: TAH; Open hysterectomy
  Arms: 1
Procedure: Total Laparoscopic Hysterectomy — The technique of total laparoscopic hysterectomy (TLH), utilising the McCartney tube, has been developed by Anthony J. McCartney over the last 10 years. It allows the completion of the hysterectomy entirely laparoscopically, without the need for additional vaginal surgery.
  Other Names: Keyhole hysterectomy
  Arms: 2

SUMMARY:
The primary objective of this study is to assess disease-free survival at 4.5 years postoperatively for women with apparent Stage 1 endometrial cancer, comparing patients who are randomised to receive Total Laparoscopic Hysterectomy (TLH) and patients who are randomised to receive Total Abdominal Hysterectomy (TAH).

DETAILED DESCRIPTION:
This phase III international, multicenter, open-label, randomized clinical trial is an equivalence study with the hypothesis is that Total Laparoscopic Hysterectomy (TLH) is associated with equivalent disease-free survival when compared to the standard treatment of Total Abdominal Hysterectomy (TAH) for women with apparent Stage I endometrial cancer.

The secondary hypotheses are:

* TLH is associated with equivalent or improved Quality of Life (QoL) at 6 months;
* TLH is associated with reduced treatment-related morbidity;
* TLH is associated with shorter hospital stay;
* TLH is associated with less analgesic consumption;
* TLH is cost effective;
* TLH is associated with improved pelvic floor function.

ELIGIBILITY:
Inclusion Criteria:

Patients who may be included for this study must have the following:

* Histologically confirmed primary endometrioid adenocarcinoma of the endometrium;
* Clinical stage I disease;
* ECOG Performance status of 0-1;
* Signed written informed consent;
* Females, aged 18 years or older.

Exclusion Criteria:

Patients will be excluded from participating from the study if they have any of the following:

* Other histologic type than endometrioid adenocarcinoma of the endometrium;
* Clinically advanced disease (stages II-IV);
* Uterine size larger than 10 weeks gestation;
* Estimated life expectancy of less than 6 months;
* Enlarged aortic lymph nodes;
* Unfit for Surgery: serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator);
* Patient compliance and geographic proximity that does not allow adequate follow-up;
* Unfit to complete QoL measurements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 760 (Actual)
Dates: Start 2005-10 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Disease free survival | 4.5 years from surgery

SECONDARY OUTCOMES:
Intra/Peri/Post-operative and long-term morbidity | 30 days from surgery
Patterns of recurrence | 4.5 years from surgery
Pain and analgesia | 1 week, 1 month, 3 months and 6 months postoperative.
Quality of Life | Measured at baseline, then again 1 week, 6 weeks, 3 months and 6 months postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Obermair, Principal Investigator — Queensland Centre for Gynaecological Cancer
Locations (23):
- Australia (19):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - John Hunter Hospital, New Lambton, New South Wales
  - Newcastle Private Hospital, New Lambton Heights, New South Wales
  - Royal Hospital for Women, Randwick, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - The Wesley Hospital, Auchenflower, Queensland
  - Greenslopes Private Hospital, Greenslopes, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Mater Adult Public Hospital, South Brisbane, Queensland
  - Mater Misericordiae Hospital Townsville, Townsville, Queensland
  - Townsville Hospital, Townsville, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Royal Women's Hospital, Carlton, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Cabrini Health, Malvern, Victoria
  - King Edward Memorial Hospital for Women, Perth, Western Australia
  - St John of God Hospital, Subiaco, Western Australia
- Queen Mary Hospital, Pok Fu Lam, Hong Kong
- New Zealand (2):
  - Christchurch Women's Hospital, Christchurch, Canterbury
  - Oxford Clinic Women's Health, Christchurch
- Royal Infirmary of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Janda M, Gebski V, Forder P, Jackson D, Williams G, Obermair A; LACE Trial Committee. Total laparoscopic versus open surgery for stage 1 endometrial cancer: the LACE randomized controlled trial. Contemp Clin Trials. 2006 Aug;27(4):353-63. doi: 10.1016/j.cct.2006.03.004. Epub 2006 May 5. PMID 16678497
- [Derived] Gebski V, Obermair A, Janda M. Toward Incorporating Health-Related Quality of Life as Coprimary End Points in Clinical Trials: Time to Achieve Clinical Important Differences and QoL Profiles. J Clin Oncol. 2022 Jul 20;40(21):2378-2388. doi: 10.1200/JCO.21.02750. Epub 2022 May 16. PMID 35576502
- [Derived] Janda M, Gebski V, Davies LC, Forder P, Brand A, Hogg R, Jobling TW, Land R, Manolitsas T, Nascimento M, Neesham D, Nicklin JL, Oehler MK, Otton G, Perrin L, Salfinger S, Hammond I, Leung Y, Sykes P, Ngan H, Garrett A, Laney M, Ng TY, Tam K, Chan K, Wrede CD, Pather S, Simcock B, Farrell R, Robertson G, Walker G, Armfield NR, Graves N, McCartney AJ, Obermair A. Effect of Total Laparoscopic Hysterectomy vs Total Abdominal Hysterectomy on Disease-Free Survival Among Women With Stage I Endometrial Cancer: A Randomized Clinical Trial. JAMA. 2017 Mar 28;317(12):1224-1233. doi: 10.1001/jama.2017.2068. PMID 28350928
- [Derived] Belavy D, Janda M, Baker J, Obermair A. Epidural analgesia is associated with an increased incidence of postoperative complications in patients requiring an abdominal hysterectomy for early stage endometrial cancer. Gynecol Oncol. 2013 Nov;131(2):423-9. doi: 10.1016/j.ygyno.2013.08.027. Epub 2013 Sep 3. PMID 24007947
- [Derived] Kondalsamy-Chennakesavan S, Janda M, Gebski V, Baker J, Brand A, Hogg R, Jobling TW, Land R, Manolitsas T, Nascimento M, Neesham D, Nicklin JL, Oehler MK, Otton G, Perrin L, Salfinger S, Hammond I, Leung Y, Sykes P, Ngan H, Garrett A, Laney M, Ng TY, Tam K, Chan K, Wrede DH, Pather S, Simcock B, Farrell R, Robertson G, Walker G, McCartney A, Obermair A. Risk factors to predict the incidence of surgical adverse events following open or laparoscopic surgery for apparent early stage endometrial cancer: results from a randomised controlled trial. Eur J Cancer. 2012 Sep;48(14):2155-62. doi: 10.1016/j.ejca.2012.03.013. Epub 2012 Apr 12. PMID 22503396
- [Derived] Janda M, Gebski V, Brand A, Hogg R, Jobling TW, Land R, Manolitsas T, McCartney A, Nascimento M, Neesham D, Nicklin JL, Oehler MK, Otton G, Perrin L, Salfinger S, Hammond I, Leung Y, Walsh T, Sykes P, Ngan H, Garrett A, Laney M, Ng TY, Tam K, Chan K, Wrede CD, Pather S, Simcock B, Farrell R, Obermair A. Quality of life after total laparoscopic hysterectomy versus total abdominal hysterectomy for stage I endometrial cancer (LACE): a randomised trial. Lancet Oncol. 2010 Aug;11(8):772-80. doi: 10.1016/S1470-2045(10)70145-5. Epub 2010 Jul 16. PMID 20638899
- See also: Gynaecological Oncology website — http://www.obermair.info
- See also: QCGC Research — http://www.gyncan.org/